CLINICAL TRIAL: NCT06949709
Title: Effects of Fasted- Versus Fed-exercise on Glucose, Lipid and Blood Pressure Responses in Physically Active Adults
Brief Title: Effects of Fasted- Versus Fed-exercise on Metabolic Health in Physically Active Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202310HM014-2
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Glucose Levels; Lipid Profile; Substrate Oxidation; Blood Pressure; Insulin Sensitivity
Keywords: Fasted-exercise; Glucose control; Lipid oxidation
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted-exercise (Experimental): Breakfast intake before 30 min walking
  Interventions: Behavioral: Fasted-exercise
- Fed-exercise (Experimental): 30 min walking before breakfast intake
  Interventions: Behavioral: Fed-exercise

INTERVENTIONS:
Behavioral: Fasted-exercise — Breakfast intake before 30 min brisk walking on a treadmill
  Arms: Fasted-exercise
Behavioral: Fed-exercise — 30 min brisk walking on a treadmill before breakfast intake
  Arms: Fed-exercise

SUMMARY:
The purpose of this study is to investigate whether the sequence meal and exercise (exercise before meal or exercise after meal) affects the postprandial metabolism.

DETAILED DESCRIPTION:
In the 48 h prior to each main trial, participants were asked to refrain from performing any strenuous physical activity and from consuming alcohol/caffeine for 24 h prior to the main trials. A dietary record was completed 24 h before the first main trial and participants were asked to replicate this diet prior to their second main trial.

On main trial days, participants arrived at the laboratory between 8-9 am following a 12-hour fast. The entire experiment lasted a total of 375 minutes. After anthropometric measurements, participants rested on a bed for 20 minutes, during which expired gas samples were collected. During the initial 60 minutes, participants then either consumed a meal before exercise (ME) or after exercise (EM). Participants were asked to finish their breakfast within 10 minutes. In both the ME and EM treatments, participants walked on the treadmill at 6 km/h (for females) and 6.4 km/h (for males) for 30 minutes. Expired gas samples were collected during this time, heart rate (HR) was monitored every 5 minutes and ratings of perceived exertion (RPE) were recorded every 10 minutes. After a 2-hour rest, lunch was provided and consumed within 15 minutes. Participants then underwent a 3-hour observation period during the postprandial phase.

Measurement:

Blood pressure was measured every 30 minutes during the experiment using the OMRON HEM-7320 blood pressure monitor (OMRON Co., Ltd., Japan). Three measurements of blood pressure and pulse were taken, and these values were averaged to ensure that the two readings were within 5 mmHg of each other. If the two readings differed by more than 5 mmHg, additional readings were taken until the outlying measurement was excluded. Blood pressure and pulse were assessed with the individual in a semi-sitting position on the bed, ensuring the arm was properly positioned.

Blood samples were taken at 0, 30, 60, 75, 90, 105, 120, 150, 180, 195, 210, 225, 240, 255, 285, 315, 345, and 375 minutes. The samples were appropriately processed, frozen, and stored in the Exercise Physiology Laboratory refrigerator at the Gongguan Campus of National Taiwan Normal University.

Gas sampling was conducted five times during the experiment. Samples were collected upon arrival at the laboratory, during exercise, one hour after breakfast or exercise, one hour after lunch, and two hours after lunch to determine resting metabolic rate (RMR) and energy expenditure using substrate oxidation.

Subjective self-assessments of appetite and mood were taken at 0, 30, 60, 120, 180, 195, 255, 315, and 375 minutes using a Visual Analog Scale (VAS) ranging from 0 to 100.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 45 years
2. Regular walking habit of at least 7500 steps per day
3. Engage in continuous walking for at least 20 minutes on 2 or more days per week
4. Body Mass Index (BMI) ranging from 18.5 to 27 kg/m2
5. No habits of heavy drinking or smoking, or have quit smoking for at least 6 months
6. Absence of diabetes, cardiovascular, or metabolic-related disorders
7. Not currently taking prescription drugs, over-the-counter medications, or other supplements that may affect blood sugar, blood pressure, or metabolic changes
8. No current sports injuries or medical advice against exercise
9. No significant weight fluctuations in the past three months (within ±3% of usual body weight)
10. Not experiencing shift work or travel across time zones within the past six months
11. No current plans to change lifestyle habits and willing to adhere to the requirements of the study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Glucose responses | 375 minutes
  Changes in glucose concentrations between trials
Insulin responses | 375 minutes
  Changes in insulin concentrations between trials

SECONDARY OUTCOMES:
Triacylglycerol responses | 375 minutes
  Changes in Triacylglycerol concentrations between trials
Blood pressure | 375 minutes
  Changes in blood pressure (e.g., diastolic and systolic blood pressure) between trials
Heart rate variability (HRV) | 375 minutes
  Changes in heart rate variability between trials
Cognitive function | 375 minutes
  Changes in cognitive function (e.g., Accuracy and reaction time) between trials
Visual Analog Scales (VAS) | 375 minutes
  Changes in VAS (e.g, appetite and mood) between trials

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan